CLINICAL TRIAL: NCT03429322
Title: Testing an Integrated Medical and Resource Facilitation Intervention After Traumatic Brain Injury: A Community-based Pragmatic Clinical Trial
Brief Title: Medical and Resource Facilitation Intervention After Traumatic Brain Injury
Acronym: MRFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Minnesota Brain Injury Alliance (Unknown); Minnesota Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-009300; 90DPTB0012-01-00 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2018-01-31; First posted 2018-02-12 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Brain Injuries, Traumatic; Family; Physician's Role
Keywords: traumatic brain injury; pragmatic clinical trial; telemedicine; cost
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Community-based randomized pragmatic clinical trial of a complex behavioral intervention delivered remotely
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Care and Resource Facilitation (Experimental): All intervention components will be delivered remotely: there will be no face-to-face interaction with the participants. The intervention is comprised of the clinical, educational, and supportive services of Mayo's Brain Rehabilitation Clinic integrated with the MN BIA RF program.
  Interventions: Behavioral: Medical Care and Resource Facilitation
- Usual care (Active Comparator): Individuals with TBI, their family members and PCPs assigned to the usual care group will receive care and provide services as usual in their communities. Individuals with TBI assigned to the usual care group will receive RF as routinely provided by MN BIA.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Medical Care and Resource Facilitation — The intervention expands on an established web-based platform and uses other information and communication technology (ICT) devices, incorporating synchronous direct clinical care and asynchronous intervention. Participants will use their own devices and internet access for any and all interactions with Mayo Clinic providers. The specific ICT modes used and services provided to interact with participants will be determined by clinical need, individual preference, and technological capacity.
  Arms: Medical Care and Resource Facilitation
Other: Usual Care — Participants will receive and provide usual and customary care in their communities.
  Arms: Usual care

SUMMARY:
Mayo Clinic's Traumatic Brain Injury (TBI) Model System Center (TBIMSC) will capitalize on longstanding collaborations with the non-profit Minnesota Brain Injury Alliance (MN BIA) and Minnesota Department of Health (MDH) to test a new way of delivering medical and social services. This trial will address chronic unmet needs expressed by individuals with TBI and their families in the U.S. pertaining to the ineffective connection to specialized medical and community resources in the transition from hospital to community-based care, limited access to TBI experts, and lack of primary care provider (PCP) knowledge about the complex needs of individuals with TBI. Target populations for this study are: 1) individuals with TBI eligible for MN BIA provided Resource Facilitation (RF), 2) their families, and 3) their PCPs.

This clinical trial will use a theory-driven complex behavioral intervention that integrates the medical-rehabilitation, therapy, and TBI expertise of Mayo's Brain Rehabilitation Clinic (BRC) with MN BIA's highly developed RF program (a free two-year telephone support service offering assistance in navigating life after brain injury). Mayo Clinic's medical-rehabilitation expertise will be integrated with RF services to deliver direct clinical care remotely using telemedicine and other information and communication technology to test whether outcomes over time are better in a group receiving this model of care compared to a group that receives usual care in their communities.

Costs between usual care and intervention groups will be compared in collaboration with the MDH. The overarching goal is development of a replicable, sustainable, and cost effective model of telemedicine care that integrates TBIMS Centers and BIAs nationwide and builds TBI expertise and capacity among PCPs.

DETAILED DESCRIPTION:
This Integrated Medical and Resource Facilitation Intervention (MRFI) trial will address: 1) The ineffective connection of individuals with traumatic brain injury (TBI) and their families to specialized medical and community resources after hospital-based care; 2) Limited access to TBI experts, and; 3) A lack of knowledge by primary care providers (PCP) about the complex needs of individuals with TBI.

This clinical trial will test a theory-driven complex behavioral intervention that integrates the medical and TBI expertise of Mayo's Brain Rehabilitation Clinic (BRC) with Minnesota Brain Injury Alliance's (MN BIA) highly developed Resource Facilitation (RF) program.

The target populations for the proposed study are: 1) Individuals with TBI eligible for MN BIA RF services; 2) Their families or caregivers; and 3) Their PCPs.

This research uses a community-based pragmatic clinical trial (PCT) to test a complex behavioral intervention. A PCT: 1) Compares multiple clinically relevant interventions rather than comparing an intervention of interest against a placebo or control condition; 2) Includes a heterogeneous population of participants in multiple experimental settings as opposed to a narrowly controlled homogeneous sample in practice settings of a single kind; and 3) Measures a broad range of health care outcomes.

The active elements in the proposed trial define a 'complex behavioral intervention'. The intervention's integrated MRFI model of care consists of: multiple components within the experimental and control interventions that interact; multiple and complex behaviors associated with those delivering and receiving the intervention; multiple target populations; multiple outcome measurements; and, adapting the intervention based on need and context.

At trial's end, the investigators will estimate the difference in the use of health care resources between individuals with TBI who receive the intervention versus those who receive usual care, by completing a cost-effectiveness analysis. True success of a clinical intervention is achieved when its benefits are realized at a similar or diminished cost compared to an alternative treatment.

Specific Aims Specific Aim 1: To assess the effectiveness of a medical/RF intervention provided remotely in improving participation outcomes of individuals with TBI when compared to a similar group receiving usual care.

Hypothesis 1: Participants receiving the trial intervention will show greater improvement in participation outcomes when compared to those receiving usual care.

Specific Aim 2: To test for the differences in caregiver burden and quality of life in the families of individuals with TBI involved in each arm of this trial.

Hypothesis 2: The family members of individuals with TBI receiving the trial intervention will report lower caregiver burden and higher quality of life when compared to family members of individuals with TBI receiving usual care.

Specific Aim 3: To measure differences in efficacy and mastery among PCPs in caring for individuals with TBI.

Hypothesis 3: PCPs for individuals with TBI receiving the trial intervention will report higher self-efficacy and mastery, when compared to providers for individuals with TBI receiving usual care.

Specific Aim 4: To compare the cost-effectiveness of the integrated service intervention arm of the trial with the usual care arm.

Hypothesis 4: Cost-effectiveness will be the same or less overall for individuals with TBI receiving the trial intervention when adjusted for covariates compared to those individuals receiving usual care.

Methods Sample Minnesota has statutory authority to identify individuals discharged from hospitals with TBI for epidemiological surveillance and to connect them with the MN BIA to offer RF. During subsequent RF intake, the recruitment and consent process will commence with RF staff introducing the study. A list of interested individuals will be securely submitted to the Mayo Research Coordinator; these individuals will then be contacted for consent and randomized. If the individual with TBI is unable to consent based on a cognitive screen, their legal representative will be approached. Participants will not be required to have a family member or PCP enrolled to be eligible for the study, but will be strongly encouraged to involve both. A consented participant's family and PCP will be contacted for consent as research participants. They will be assigned to the same group as the individual with TBI. Randomization to ensure representation of known prognostic factors where age (≤65 and >65), gender, and residence (rural or urban) will be used as stratification factors, with treatment assignment balanced in blocks of 4. Because a simple random scheme may limit enrollment of rural participants the investigators will over-sample in a ratio of 2:1 rural/urban.

Sample Size and Power Calculations For Specific Aim 1, a sample size of 500 individuals is considered desirable based on power calculations as described. By achieving this sample size a minimum difference of at least 0.25 standard deviations can be detected between groups for each continuous outcome of interest, with 80% power based on a two-sample t-test. In 2014, 3,868 people 15 years old or older were hospitalized with TBI in MN and 1,108 people with TBI received RF in MN in 2016. The investigators plan a 24-month enrollment period, so 2,216 individuals with TBI will be potentially eligible. The minimum detectable difference between the groups based on a two sample t-test will be 0.25 standard deviations. The sample size of 250 per group will have 80% power to detect a correlation of 0.18 or larger between any two continuous outcomes within the group. For an assessment of associations between group and other categorical variables, there would exist 80% power to detect a difference of 11% or larger for the presence of a categorical outcome (15% among participant with usual care versus 25% among participants receiving the study intervention) based on a Chi-square test of two proportions.

Intervention All intervention components will be delivered remotely: there will be no face-to-face interaction with the research participants. The complex intervention being tested is comprised of the clinical, educational, and supportive services of the Mayo BRC integrated with the MN BIA RF program. The specific ICT modes used to interact with intervention participants, and the specific clinical services that are provided by these modes, will be determined by clinical need, individual preference, and technological capacity.

Individuals with TBI, their family members and PCPs assigned to the usual care group will receive care and provide services as usual in their communities. Individuals with TBI assigned to the usual care group will receive RF as routinely provided by MN BIA. For individuals with TBI, their families and PCPs assigned to the intervention group, their health, social, community, education, support, resource, and care coordination needs will be assessed. Individuals with TBI assigned to the intervention group will receive RF as integrated into the intervention.

Every intervention group participant in all target populations will receive a unique combination of services. It is expected that the composition of each participant's integrated team will vary based on individual needs, preferences, and technological capacity. Ideally, all teams will include a PCP. If a PCP is not already established, the Advanced Practice Registered Nurse will help facilitate this.

The MRFI intervention expands on a previously established web-based platform and other ICT, incorporating synchronous direct clinical care (telemedicine). Other synchronous and asynchronous intervention will be delivered as needs indicate. Participants will use their own devices and internet access for any and all interactions with Mayo Clinic providers.

Data Analysis Data for continuous variables will be summarized using descriptive statistics. Frequencies and percentages will be calculated for categorical variables. Baseline characteristics and demographic variables will be compared using two sample t-test or Wilcoxon rank sum test for continuous variables and using Chi-square test or Fisher's exact test for categorical variables of interest. Associations between continuous variables within each group will be estimated using Pearson or Spearman correlation coefficient. Comparison of correlations across the groups of interests will be performed using the Fisher's r-to-z transformation, which calculates a value of z that can be applied to assess the significance of the difference between two correlation coefficients. All the statistical tests will be 2-sided with an alpha level of 0.05.

Statistical analysis for Specific Aim 1 For each individual outcome measure the investigators will first compute percent change from baseline to last follow-up measurement to account for baseline measurements. Further analysis will be performed using these percent changes. However, analyzing effectiveness using each individual measure will not provide a single p-value to measure the intervention's overall effect on participation outcomes. Therefore, the investigators will perform the analysis using a composite endpoint that will allow us to assess the global impact of the intervention using single comparisons performed as two sample t-tests or a Wilcoxon rank sum test.

All analyses will be performed on an intent-to-treat basis. If there are any baseline covariate imbalances between the groups, the investigators will perform linear regression analyses, where summed ranks for each individual will be an outcome of interest and the primary predictor variable will be group, adjusting for those covariates that had imbalances among the groups at baseline.

Statistical analysis for Specific Aims 2 and 3 The primary goal of these Aims is to measure caregiver burden and family needs, and efficacy and clinical mastery in PCPs. Percent change from baseline will be reported as mean and standard deviation or median as appropriate. Comparisons of percents between the groups assigned to intervention versus usual care will be performed using two sample t-tests or Wilcoxon rank sum test as appropriate. If there is imbalance in any baseline covariates of interest, analysis will be performed using linear regression adjusting for those covariates of interest.

Statistical analysis for Specific Aim 4 In order to assess the cost-effectiveness of the proposed intervention, the trial patients will be linked to the Minnesota All Payers Claims Database (MN-APCD) developed and maintained by MDH. Both healthcare utilization and cost outcomes will be compared between the participants in the intervention and usual care arms. Adjustments will be made to account for different payment levels between governmental and commercial payers. Descriptive statistics of these outcomes including mean, median, and standard deviation will be provided. If any difference between the intervention and usual care groups in terms of their baseline characteristics is observed, multivariate adjustments will be conducted; due to expected skewness of underlying distribution, utilization outcomes will be analyzed using count regression (e.g., negative binomial regression) while cost will be analyzed using generalized linear modeling with gamma distribution for cost, and logarithmic link. In order to meet the confidentiality terms of the data submitters to MN-APCD, trial participants' records will be matched by applying the same MN algorithms to generate the hashed identifiers used to link claims for the same person through the following set of identifiers: name (first, middle, and last name), 5-digit zip code, age, gender, and date of birth. To carry out this linkage and avoid the possibility of participant re-identification, the creation of the analytic dataset from MN-APCD and subsequent analyses will be conducted by the MDH staff. The match rate of the trial participants to the MN-APCD will be reported.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Diagnosis of traumatic brain injury
* Minnesota resident
* Access to at least a telephone
* Functional English speaker
* Eligible for MN BIA Resource Facilitation participant

Exclusion criteria:

* Age < 18 years
* Diagnosis of acquired brain disorder other than traumatic brain injury
* No telephone or on-line/internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Change in Mayo-Portland Participation Index (M2PI) | Collected 3 times: enrollment, midpoint (6 months), and study end (18 months)
  A primary participation assessment and outcome measure for phone follow-up
Change in Traumatic Brain Injury-Quality of Life (TBI-QOL) | Collected 3 times: enrollment, midpoint (6 months), and study end (18 months)
  Measures health-related patient-reported quality of life measurement specific to TBI
Change in Participation Assessment with Recombined Tools-Objective (PART-O) | Collected 3 times: enrollment, midpoint (6 months), and study end (18 months)
  Measures long-term outcomes and function at the societal level

SECONDARY OUTCOMES:
Change in Vocational Independence Scale | Collected 3 times: enrollment, midpoint (6 months), and study end (18 months)
  Quantifies degree of vocational independence: 5-point ordinal scale which quantifies the degree of vocational independence, where level 1 is unemployed and level 5 is independent engagement in community-based work (at least 15 hours per week) without external supports.
Change in Telemedicine Perception Questionnaire (TMP-Q) | Collected 3 times: enrollment, midpoint (6 months), and study end (18 months)
  Assesses impressions of the risks and benefits of home tele-care
EQ-5D™ | Assessed at study end (18 months)
  A measure of health outcome to be used in determining cost-effectiveness
Change in Zarit Burden Inventory (ZBI) | Collected 3 times: enrollment, midpoint (6 months), and study end (18 months)
  Caregiver burden self-report measure
Change in Family Needs Questionnaire (FNQ) | Collected 3 times: enrollment, midpoint (6 months), and study end (18 months)
  Assesses diverse family needs
Change in Clinical Satisfaction and Competency Rating Scale (CSCRS) | Collected 3 times: enrollment, midpoint (6 months), and study end (18 months)
  Measures provider efficacy and mastery in caring for individuals with TBI: a 7 question format with each question rated in a 5-point scale with 1=disagree and 5=agree. The highest score of 35 indicates the best satisfaction and competency and the lowest score of 7 indicates the worst clinical satisfaction and competency.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Esterov, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials